CLINICAL TRIAL: NCT00468832
Title: Longitudinal Study of the Relationship Between Impairment, Activity Limitation, Participation and Quality of Life in Persons With Confirmed Duchenne Muscular Dystrophy (DMD)
Brief Title: Longitudinal Study of the Natural History of Duchenne Muscular Dystrophy (DMD)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Cooperative International Neuromuscular Research Group (Network)
Collaborators: U.S. Department of Education (U.S. Federal Agency); National Institutes of Health (NIH) (NIH); United States Department of Defense (U.S. Federal Agency); Parent Project Muscular Dystrophy (Other)
Responsible Party: Sponsor
Other Study IDs: UCD0305
Record Dates: First submitted 2007-05-01; First posted 2007-05-03 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples are being collected for single-nucleotide polymorphism, Genome-wide Association Study, and biomarker analyses.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Ongoing Duchenne Muscular Dystrophy (DMD) Cohort: 340 patients currently enrolled participants with DMD.
- New Young Duchenne Muscular Dystrophy (DMD) Cohort: Additional 100 confirmed DMD participants aged 4-7 years old to be recruited.
- Typically Developing Control Cohort: Up to 370 typically developing male children and adults aged 6-30 years old to be recruited.

SUMMARY:
The purpose of this study is to establish the largest long-term assessment of people with Duchenne muscular dystrophy (DMD). In this study, the investigators associated with the Cooperative International Neuromuscular Research Group CINRG) will take a detailed look (for a minimum of eight years) at DMD participant's physical abilities, the medical problems they experience, and how they use health care services. Physical abilities will be compared to a group of healthy controls.

The second purpose of this study is to find out whether small, normal differences in the genetic makeup of people with DMD (called "single nucleotide polymorphisms" or "SNPs") affect how their disease progresses and relates to muscle strength/size and steroid response.

The third purpose of this study is to study genetic variations associated with DMD.

The final purpose of this study is to determine whether certain biomarkers are present in people with DMD and not in healthy controls.

DETAILED DESCRIPTION:
Phenotyping Study Aims

Aim 1: Longitudinally assess body function and body structure (impairment) through the measurement of anthropometrics, muscle strength and pulmonary function in subjects with DMD through the multicenter CINRG network.

Aim 2: Longitudinally assess activity limitations in subjects with DMD through CINRG with timed motor performance, burden of care, and functional status.

Aim 3: Longitudinally assess secondary conditions in subjects with DMD, and relative risks of developing those conditions based on exposure to preventive interventions.

Aim 4: Longitudinally assess participation, life satisfaction, service utilization and health-related quality of life in subjects with DMD.

Aim 5: Determine appropriate outcome measurements for impairment, activities (activity limitations), participation and quality of life to determine the effect of prednisone and other therapeutic interventions on these factors.

Aim 6: Using the most robust impairment, activity, participation and quality of life outcome measures, determine the sample size, power and statistical methods for the analysis of the effect size for future planned randomized-controlled rehabilitation interventions in DMD.

Aim 7: Examine the associations between interventions and incidence and severity of secondary conditions, achievement of disease milestones and measures of motor function and mobility.

Aim 8: To assess the validity and responsiveness of novel clinical outcome measures in DMD, including the 6-minute walk test (6MWT), the 9-hole peg test (9-HPT) Egen Klassification Scale(EK), the North Star Ambulatory Assessment (NSAA), and quantitative key and pinch grip strength testing.

Aim 9: To assess the reliability, validity and responsiveness of novel patient-reported outcome(PRO) measures in DMD, including the NeuroQOL and PedsQL Neuromuscular Module.

Aim 10: To assess the clinical meaningfulness of novel objective clinical outcome measures by assessing their ability to predict milestones of loss of ability to stand from supine, to stand from a seated position, to climb stairs, to ambulate independently and to raise a hand to the mouth.

AIM 11: To determine the impact of development and growth on outcome measure performance,we will assess physical function on a group of healthy, typically developing male children and adults between 6 and 30 years of age for outcome measures of motor function and strength including the9-HPT, 6MWT, NSAA, timed function tests and quantitative muscle strength (QMT). Test results from this cohort will be used to develop initial percent predicted for age values for these assessments.

SNP Genotyping Study Aim

Our goal of the proposed study is to define polygenic modifiers of disease progression, and also response to treatment with glucocorticoids (prednisone and deflazacort). The most common type of human genetic variation is the single-nucleotide polymorphism (SNP, a base position at which two alternative bases occur at an appreciable frequency (>1%) in the population. SNPs are 90% of variation in the human genome. SNPs occur on the average of 1 per 1000 to 2000 bp throughout the 3.2 billion bp of the human genome while coding region SNPs (cSNPs) occur on the average of 1 per 346 bp.

Genome-wide Association Study Aim

Our goal of the proposed study is to isolate genomic DNA and find possible correlations of clinical phenotypes with gene loci associated with mild vs. severe clinical presentation, progression, or response to steroids.

Serum Biomarkers Study Aim

Our goal is to discover and validate sensitive and specific serum biomarkers for DMD.

ELIGIBILITY:
DMD Subject Inclusion Criteria

* Affected subjects must be male and between the ages of 2 and 30
* Affected subjects between the ages of 2 and 4 must have a diagnosis of DMD confirmed by at least one the following OR have an older male sibling that meet at least one of the following criteria:

  * Dystrophin immunofluorescence and/or immunoblot showing complete dystrophin deficiency, and clinical picture consistent with typical Duchenne dystrophy OR
  * Gene deletion test positive (missing one or more exons) in the central rod domain exons 25-60) of dystrophin, where reading frame can be predicted as 'out-of-frame',and clinical picture consistent with typical Duchenne dystrophy.
  * Complete dystrophin gene sequencing showing an alteration (point mutation, duplication, other) that is expected to preclude production of the dystrophin protein(i.e. nonsense mutation, deletion/duplication leading to a downstream stop codon),with a typical clinical picture of DMD.
* Affected subjects between the ages of 5 and 30 must either fulfill the above criteria OR show evidence of a dystrophinopathy and clinical picture consistent with Duchenne Muscular Dystrophy

  * Participants who have documented clinical symptoms referable to a dystrophinopathy and direct support of the diagnosis by either (1) a positive DNA analysis for dystrophin mutation, (2) a muscle biopsy demonstrating abnormal dystrophin, or (3) an elevated CK (>5X normal), and X-linked pedigree and an affected family member who meets either criterion (1) or (2) as described above.

NOTE: Determination of the appropriate clinical symptoms consistent with DMD will generally be the responsibility of the clinician. At a minimum this will include progressive loss of function, with additional consideration for other clinical features such as a characteristic gait, a positive Gower sign and calf pseudohypertrophy. When immunostaining of muscle biopsy is used to determining case definition, the clinical reviewer (site PI) should confirm that appropriate testing has ruled out a secondary deficiency of dystrophin. Affected subjects that do not exhibit the above symptoms consistent with DMD should be excluded.

o Muscle weakness prevalent by 5 years of age

- Non-affected adult subjects must be Parent(s) or legal guardian(s) of an eligible affected subject.

DMD Serum Biomarker Inclusion Criteria

* Participants must meet eligibility criteria for the DMD phenotyping portion of this study
* For the GC-treatment response cohort, participants must initiate GC treatment within the first year of study participation (i.e. between their first study visit and their one year follow-up visit)

DMD Subject Exclusion Criteria

For those subjects that confirm DMD diagnosis through a clinical picture consistent with DMD

* Steroid-naïve subjects ambulating past the 13th birthday
* Steroid users ambulating past the 16th birthday
* Subjects/families who are unwilling or unable to comply with the protocol study procedures or visits

Controls Subject Inclusion Criteria

* Male sex
* Age 6-30 years
* Able to comply with functional testing instructions

Control Serum Biomarker Inclusion criteria

* Participants must be male
* Participants must be free of DMD, other neuromuscular disease, or other significant concomitant illness
* Participant must be free of glucocorticoid therapy

Control Subject Exclusion Criteria

* Musculoskeletal disease
* Musculoskeletal injury within 6 months of enrollment
* Other concomitant illness that precludes functional testing in the judgment of the investigator or clinical evaluator
* Completion of enrollment for age cohort

Ages: 2 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The incidence of DMD is considered equal across racial and ethnic groups. At the start of the CINRG program, it was assumed by investigators that the aggregate subject populations of the participating US sites should closely mirror the racial and ethnic distribution of the US population.
  DMD is an X-linked recessive disease affecting only males. However, female carriers of the disease can be symptomatic due to skewed X-inactivation, a secondary genetic event. We have opted to study the most commonly affected population, males, to ensure subject homogeneity. As such, there are no outreach programs planned for women in this study.
Sampling Method: Non-Probability Sample
Enrollment: 551 (Actual)
Dates: Start 2005-12; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Strength and function | Collected at yearly visits
  These assessments include:
  * Quantitative muscle testing
  * Manual muscle testing
  * Pulmonary function testing
  * Functional evaluations (nine hole peg, six minute walk, North Star ambulatory assessment, Brooke and Vignos scales, Egen Klassification (EK) scale, and range of motion).
Quality of life | Collected at yearly visits
  These questionnaires include:
  * Pediatric Quality of Life Inventory (PedsQL)
  * Pediatric Orthopaedic Functional Health Questionnaire of the Pediatric Orthopaedic Society of North America (POSNA)
  * World Health Organization Quality of Life Assessment - Brief (WHO QOL Brief)
  * Pediatrics and Adult Neuromuscular module Quality of Life (NeuroQOL)
  * Review of Systems
Medical history assessment | Collected at yearly visits
  Outcomes on ambulation status, medication history, hospitalizations, surgeries, nutrition, fractures, and cardiac tests.

SECONDARY OUTCOMES:
Biomarkers and genetic modifiers | Collected either once at any visit or each visit
  Genotyping and Serum Biomarkers include blood/saliva collection for:
  * Blood collection for Genome Wide Association Study (GWAS) analysis (one time sample, any visit)
  * Blood or saliva collection for SNP sample (one time sample, any visit)
  * Blood collection for biomarker analysis (collected at each visit)

CONTACTS AND LOCATIONS:
Overall Officials: Craig McDonald, MD, Study Chair — University of California, Davis
Locations (21):
- United States (11):
  - University of California, Davis, Sacramento, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of of Florida, Gainesville, Florida
  - Lurie Children's Hospial, Chicago, Illinois
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University, St. Louis, St Louis, Missouri
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke Children's Hospital, Durham, North Carolina
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - University of Tennessee, Memphis, Tennessee
  - Children's Hospital of Virginia, Richmond, Virginia
- Fundacion Favaloro, Buenos Aires, Argentina
- Australia (2):
  - The Children's Hospital at Westmead, Sydney, New South Wales
  - Royal Children's Hospital, Melbourne, Victoria
- Canada (3):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Holland Bloorview Kids Rehab Hospital, Toronto, Ontario
- Apollo Hospitals, Chennai, India
- Schneider Children's Medical Center of Israel, Petach Tikvah, Israel
- NEMO, Milan, Italy
- Queen Silvia Children's Hospital, Gothenburg, Sweden

REFERENCES:
- [Derived] Thangarajh M, Spurney CF, Gordish-Dressman H, Clemens PR, Hoffman EP, McDonald CM, Henricson EK; CINRG Investigators. Neurodevelopmental Needs in Young Boys with Duchenne Muscular Dystrophy (DMD): Observations from the Cooperative International Neuromuscular Research Group (CINRG) DMD Natural History Study (DNHS). PLoS Curr. 2018 Oct 17;10:ecurrents.md.4cdeb6970e54034db2bc3dfa54b4d987. doi: 10.1371/currents.md.4cdeb6970e54034db2bc3dfa54b4d987. PMID 30443431
- [Derived] McDonald CM, Henricson EK, Abresch RT, Duong T, Joyce NC, Hu F, Clemens PR, Hoffman EP, Cnaan A, Gordish-Dressman H; CINRG Investigators. Long-term effects of glucocorticoids on function, quality of life, and survival in patients with Duchenne muscular dystrophy: a prospective cohort study. Lancet. 2018 Feb 3;391(10119):451-461. doi: 10.1016/S0140-6736(17)32160-8. Epub 2017 Nov 22. PMID 29174484
- See also: CINRG Website — http://www.cinrgresearch.org